CLINICAL TRIAL: NCT01898767
Title: Production of Eicosanoid Lipids by Airway Cells During Infection With Human Rhinoviruses: An In Vitro Model System to Study the Mechanisms of Asthma Exacerbation Resolution
Brief Title: Eicosanoid Lipids by Airway Cells During Infection With Human Rhinoviruses
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2013-0935; 1R01HL115118-01A1 (NIH)
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Asthma
Keywords: mild; asthma; allergic
MeSH Terms: conditions — Asthma; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, DNA, RNA, bronchoalveolar lavage, bronchial brushings
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Mild asthma: Diagnosis of mild asthma as defined by pre-albuterol forced expiratory volume in the first second (FEV1) of >70% predicted.

SUMMARY:
The long-range goal of this protocol is to more completely understand the risks and the pathophysiology of asthma exacerbations, in order to develop prevention strategies and/or expedite a return to complete control of baseline asthma symptoms.

DETAILED DESCRIPTION:
Theinvestigators and others have shown that airway epithelial cell infection with human rhinovirus (HRV) is a major risk factor for subsequent exacerbation. Additionally, the investigators have shown that the nucleotide receptor, P2X7, is an important host factor in the prevention of exacerbations, and have data to suggest that this may occur at the level of the alveolar macrophage. Alveolar macrophages facilitate the resolution of inflammation in part by generating eicosanoid metabolites of arachidonic acid including prostaglandin E2 (PGE2) and lipoxin A4 (LXA4). Patients with severe asthma have a reduced capacity to generate PGE2 and LXA4 when compared to those with non-severe asthma, despite alveolar macrophage expression of two of the key enzymes involved in their production. These and other data suggest that pro-resolving eicosanoid metabolism is most efficient when airway epithelial cells are in communication with alveolar macrophages, and that these pathways may be defective in patients with severe asthma. Moreover, inoculation experiments with human rhinovirus (HRV) demonstrate that alveolar macrophages express cox-2 during resolution. These and other data have led to the central hypothesis that transcellular generation of PGE2 and lipoxins is regulated by P2X7-induced cox-2 expression in alveolar macrophages, and that this process facilitates resolution of an HRV-triggered exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* Diagnosis of mild asthma
* Pre-albuterol forced expiratory volume in the first second (FEV1) of >70% predicted.
* Confirmation of asthma diagnosis by either an improvement in FEV1 after four puffs of albuterol by ≥ 12%, or a decline in FEV1 by ≥ 20% after a graded challenge with inhaled methacholine with a provocative concentration causing a 20% fall ≤ 8 mg/mL
* Documented negative Tuberculin skin test (PPD) within the last 12 months or a medical history that is consistent with a low probability of exposure to tuberculosis (i.e. the subject is not a health worker, has not traveled to endemic areas, and has no pre-existing medical or social risk factors for tuberculosis).
* Safety laboratory assessments within normal ranges (labs to include complete blood count with differential and platelet count, PT/INR, creatinine, ALT)
* Women of child-bearing potential (WCBP) must have a negative urine pregnancy test (urine HCG) within 48 hours of the methacholine challenge at Visit 2, within 48 hours of the bronchoscopy at Visit 3 and within 48 hrs of Visit 4. WCBP must agree to use a reliable method of birth control for the duration of the study (reliable methods of birth control can include abstinence, barrier methods, oral contraceptives, injection contraceptives or skin absorption contraceptives).
* In the opinion of the investigator, capable and willing to grant written informed consent and cooperate with study procedures and requirements.

Exclusion Criteria:

* Major health problems such as autoimmune disease, heart disease, type I and II diabetes, uncontrolled hypertension or lung diseases other than asthma. The listed health problems are definitive exclusion but decisions regarding major health problems not listed will be based upon the judgment of the investigator.
* No pre-existing chronic infectious disease.
* Any condition for which, in the opinion of the investigator, transient oxyhemoglobin desaturation is inadvisable.
* Pregnant or lactating females or has a planned pregnancy during the course of the study.
* Asthma maintenance therapy other than inhaled short acting beta-agonists within 1 month of screening. This includes but is not limited to inhaled or oral corticosteroids, long acting beta-agonists and leukotriene receptor antagonists.
* Upper or lower respiratory infection within 1 month of screening.
* Unstable asthma as indicated by self-report of increased symptoms or increased beta-agonist use over the 2 weeks preceding the screening visit.
* Current smokers (defined as smoked within the last year) or a former smoker with a history of >10 pack years.
* Morbid obesity as defined by a Body Mass Index (BMI) > 40.
* Use of an investigational drug within 30 days of entering the study
* History of noncompliance with medical regiments or subjects who are considered unreliable including those with a psychiatric history that, in the opinion of the investigator, may interfere with the conduct of study procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects with mild asthma from Madison, WI region
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2013-12-17 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-29 (Actual)

PRIMARY OUTCOMES:
Cox2 expression | One day
  P2X7 agonist-induced fold stimulation (over the media control) of cox2 expression (assessed by densitometry) in alveolar macrophages primed with conditioned medium from minor group HRV-infected epithelial cells.
BzATP-induced PGE2 | One day
  The amount of BzATP-induced PGE2 in the culture supernatants of alveolar macrophages primed with HRV-infected epithelial conditioned media
LXA4 produced by BzATP | One day
  The amount of LXA4 produced by BzATP co-treatment of HRV infected of epithelial-macrophage co-cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Loren Denlinger, MD/PhD, Principal Investigator — UW Madison
Locations (1):
- UW Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes